CLINICAL TRIAL: NCT03823729
Title: A Randomized, Open, Comparative Clinical Investigation to Show the Efficacy of a Short Time, Whole Body, Electrostatic High Voltage Application for Relief of Chronic Pain. Included in Study Can be Persons Suffering From Chronic Pain as it is Often Case With Rheumatic Disease or Traumata
Brief Title: Elosan Efficacy Study (EES)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elosan AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELO-02-17
Record Dates: First submitted 2019-01-25; First posted 2019-01-30 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Patients assigned to the Elosan group (group A) will have 8 sessions in the Elosan cabin, with an interval of 3 to 4 days between sessions. Patients assigned to the control group (group B) will have no treatment except for the continuation of their prescribed pain medication and pain therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elosan Cabin (Experimental): Treatment with Elosan cabin
  Interventions: Device: Elosan Cabin
- No Treatment (No Intervention): Continuation of taking pain medication as prescribed before study start.

INTERVENTIONS:
Device: Elosan Cabin — The Elosan Cabin is a closed, electrically insulated, biocompatible cabin for the short-term application of electrostatic high voltage. Patients assigned to the Group A will have 8 sessions in the Elosan cabin, with an interval of 3 to 4 days between sessions.
  Arms: Elosan Cabin

SUMMARY:
The "Elosan Cabin" is a closed, electrically insulated, biocompatible cabin for the short-term application of electrostatic high voltage in patients with chronic pain, especially those with rheumatic diseases. Patients assigned to the Elosan group (group A) will have 8 sessions in the Elosan cabin, with an interval of 3 to 4 days between sessions. Patients assigned to the control group (group B) will have no treatment except for the continuation of their prescribed pain medication and pain therapy.

DETAILED DESCRIPTION:
Included in the study can be all persons suffering from chronic pain, as it is often the case with rheumatic disease or traumata. The Elosan therapy to be investigated aims to treat chronic pain by applying an electrical charge to the body surface and by disruption of positive bio-feedback to restore physiological reflex relations between the periphery and the central regulation. The electric charge is created by a generator which can produce an electrostatic field. The electrical voltage is delivered to the hands via a metal handle in a closed cabin and is spread over the entire body surface.

A total number of 42 patients will be included into this trial in order to show a statistically significant reduction of pain compared to reduction of pain in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* adults, age ≥ 18 years, male or female patients
* History of pain ≥ 6 months
* Suffering from chronic pain, either reumatic pain or pain caused by traumata
* Intensity of pain rated ≥ 50 mm on VAS pain

Exclusion Criteria:

* Untreated thyroid disease
* History of seizure disorder (epilepsy)
* History of or current psychosis
* Women who are pregnant, breast feeding or intending to become pregnant
* Patients who are currently participating in other studies or have participated in other studies within the last 30 days
* Patients who have expressed their intention, or are suspected of intending, to discontinue therapy or stop therapy before the end of trial
* Patients with an electric or electronic implant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Change of Pain Intensity is being assessed by Visual Analogue Scale (VAS). | Change from Baseline Intensity of pain at 4 weeks
  Change of Pain Intensity is being assessed on a horizontal 100 mm VAS (Visual Analogue Scale) pain scale. The total range of this scale is 100 mm. Minimum score is 0 mm, Maximum score is 100 mm. The higher values represent a higher intensity of pain. The values at baseline will be compared to the values at Visit 8 and the mean of the differences will be compared between the 2 treatment arms.

SECONDARY OUTCOMES:
Change in quality of life is being assessed by SF 12 Questionnaire (The 12-Item Short Form Health Survey) | Change from Baseline at 4 weeks
  The change in quality of life (as reported by SF 12 questionnaires) from baseline to end of treatment (Day 28) will be compared between the treatment groups. The impact of the changes in summary scores (NBS: Norm-Based-Scoring) of physical health (PCS) and mental health (MCS) will be assessed by a General Linear Model (GLM) using the treatment as fixed factors and the baseline PCS and MCS as covariates, respectively.
Pain medication / pain therapy and any changes thereof shall be recorded during the study. | before and after 4 weeks of treatment
  The pain medication taken at baseline will be compared to the amount of pain medication taken at the end of treatment. Changes in pain medication will be qualified by the investigators as either being clinically relevant or not.

CONTACTS AND LOCATIONS:
Locations (3):
- Switzerland (3):
  - Polymedes Pain Center, Bad Ragaz, CH
  - Centro Ortho-Bio-Med, Roveredo, CH
  - Zentrum für Neurochirurgie Hirslanden Ostschweiz, Sankt Gallen, CH

IPD SHARING:
Plan to Share IPD: No